CLINICAL TRIAL: NCT05415384
Title: Single Center, Randomized Control Trial of Cryoablation During Surgical Stabilization of Rib Fractures
Brief Title: Randomized Control Trial, Cryoablation as an Adjunct to Surgical Stabilization of Rib Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00084611
Record Dates: First submitted 2022-06-06; First posted 2022-06-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative; Rib Fracture Multiple
Keywords: Locoregional pain; thoracotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The proposed study is a single center, prospective, randomized controlled trial evaluating the efficacy of adding cryoneurolysis for patients that meet indication for Surgical Stabilization of Rib Fractures (SSRF) and consent to surgical fixation
Who Masked: Participant
Masking Description: The study will blind patients to whether or not they underwent cryoneurolysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Surgical Stabilization of Rib Fractures plus Multimodal Pain Therapy plus CRYOABLATION (Experimental): Adding Cryoablation of levels 3-8, in addition to patients that undergo SSRF for multiple rib fractures.
  Interventions: Device: Cryoablation of Intercostal Nerves
- Surgical Stabilization of Rib Fractures plus Multimodal Pain Therapy (Active Comparator): Standard surgical treatment of patients with multiple rib fractures plus Multimodal Pain Therapy
  Interventions: Procedure: Standard surgical treatment of patients with multiple rib fractures

INTERVENTIONS:
Device: Cryoablation of Intercostal Nerves — Using Atricure device, cryoice, intercostal nerves 3-8 will be ablated in the experimental arm. This is in addition to mechanical fixation of rib fractures and multimodal systemic therapy.
  Arms: Surgical Stabilization of Rib Fractures plus Multimodal Pain Therapy plus CRYOABLATION
Procedure: Standard surgical treatment of patients with multiple rib fractures — Standard surgical treatment of patients with multiple rib fractures
  Arms: Surgical Stabilization of Rib Fractures plus Multimodal Pain Therapy

SUMMARY:
To determine if patients with intraoperative cryoablation have better analgesia results compared to the control group of Surgical Stabilization of Rib Fractures (SSRF) without cryoablation

DETAILED DESCRIPTION:
Locoregional pain control with cryoneurolysis of intercostal nerves has been employed as an adjunct for longer term pain control. Initially introduced in thoracic surgery, intercostal nerve cryoablation has demonstrated adequate pain control and substantial decrease in opioid consumption and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* The patient is admitted to the trauma service.
* The patient has multiple displaced rib fractures (≥2 ribs), offered fixation, and consents to SSRF
* The patient is not being treated for chronic pain
* The patient is >18 years of age.
* Surgery anticipated <120 hours from injury

Exclusion Criteria:

* Age < 18 years or ≥ 80 years
* Flail chest: either radiographic or clinical. Radiographic flail chest is defined on CT chest as ≥ 2 ribs each fractured in ≥ 2 places. Clinical flail is defined as visualization of a segment of chest wall with paradoxical motion on physical exam.
* Moderate or severe traumatic brain injury (Intra-cranial hemorrhage visualized on CT head with GCS at the time of consideration for enrollment < 12)
* Prior or expected emergency exploratory laparotomy during this admission
* Prior or expected emergency thoracotomy during this admission
* Prior or expected emergency craniotomy during this admission
* Spinal cord injury
* Pelvic fracture that has required, or is expected to require, operative intervention during this admission
* The patient was unable to accomplish activities of daily living independently prior to injury (e.g., dressing, bathing, preparing meals)
* The patient is incarcerated
* The patient is known to be pregnant
* Unable to perform Video Assisted Thoracoscopy (VATS) at time of SSRF due to lung isolation or previous pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Morphine Milligram Equivalents Use following Intervention | Baseline
  To determine if patients with intraoperative cryoablation have better analgesia results compared to the control group of SSRF without cryoablation.
Morphine Milligram Equivalents Use following Intervention | Day 1
  To determine if patients with intraoperative cryoablation have better analgesia results compared to the control group of SSRF without cryoablation.
Morphine Milligram Equivalents Use following Intervention | Day 30
  To determine if patients with intraoperative cryoablation have better analgesia results compared to the control group of SSRF without cryoablation.
Morphine Milligram Equivalents Use following Intervention | Day 90
  To determine if patients with intraoperative cryoablation have better analgesia results compared to the control group of SSRF without cryoablation.

SECONDARY OUTCOMES:
Number of days in Hospital Stay | Days during admission
  Hospital Length of Stay
Number of days in ICU Stay | Day 90
  ICU Length of Stay
Amount of Chest tube drainage | Day 90
  Chest tube drainage
Quality of Life Scores | Month 1 and Month 3
  Quality of Life questionnaire - Quality of life questionnaire consists of a set of survey questions that can be used to collect data related to an individual in particular and society in general on various parameters that determine their general quality of life
Number of Mortalities in hospital | Day 90
  Mortality, in hospital
Number of Readmissions | 30 day readmission rate
  Readmission
Number of Additional Thoracic Procedures | Day 7
  Additional Thoracic Procedures

CONTACTS AND LOCATIONS:
Overall Officials: Bradely W. Thomas, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No